CLINICAL TRIAL: NCT05756972
Title: A Phase II Clinical Trial to Evaluate the Efficacy and Safety of PM8002(Anti-PD-L1/VEGF) in Combination With Chemotherapy in Patients With EGFR-mutant Advanced Non-squamous NSCLC Who Have Failed to EGFR-TKI Treatment
Brief Title: A Study of PM8002 (Anti-PD-L1/VEGF) in Combination With Chemotherapy in Patients With NSCLC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Biotheus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM8002-BC010C-NSCLC-R
Record Dates: First submitted 2023-02-15; First posted 2023-03-07 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: NSCLC
MeSH Terms: interventions — Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PM8002+Chemotherapy (Experimental): Subjects will be administered with PM8002 plus pemetrexed and carboplatin via intravenously (IV) Q3W for 4 cycles, followed by PM8002 and pemetrexed until progression or for a maximum of 2 years.
  Interventions: Drug: PM8002; Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: PM8002 — IV infusion
Drug: Carboplatin — IV infusion
Drug: Pemetrexed — IV infusion

SUMMARY:
PM8002 is a bispecific antibody targeting PD-L1 and VEGF. This is a phase II study to evaluate the efficacy and safety of PM8002 in combination with pemetrexed and carboplatin in patients with EGFR-mutant locally advanced or metastatic non-squamous NSCLC who have failed to EGFR-TKI treatment.

DETAILED DESCRIPTION:
This study is a phase II, single-arm study, 64 participants were enrolled as of 6 Feb 2024, and recruitment was completed.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form before any trial-related processes.
2. Age ≥ 18 years male or female.
3. Have a histologically or cytologically confirmed stage IIIB/IIIC NSCLC that is unresectable and not fit for radical concurrent chemoradiotherapy, or metastatic non-squamous NSCLC (IV).
4. with EGFR mutation confirmed by tumor histology or cytology or hematology prior to EGFR-TKI treatment.
5. EGFR-TKI resistance, confirmed by RECIST v1.1.
6. have adequate organ function.
7. The investigator confirms at least one measurable lesion according to RECIST v1.1. A measurable lesion located in the field of previous radiation therapy or after local treatment may be selected as a target lesion if progression is confirmed.
8. The Eastern Cancer Cooperative Group (ECOG) performance score of 0 or 1.

Exclusion Criteria:

1. Squamous cell > 10%. If small cell types are present, the subject is not eligible for inclusion.
2. Have other driving gene mutations that can obtain effective treatment.
3. Have previously received systemic anti-tumor treatment other than EGFR-TKI for advanced non-squamous NSCLC.
4. Have received systemic steroid therapy or any other form of immunosuppressive therapy within 14 days prior to the first dose of study drugs.
5. Have received EGFR-TKI treatment, within 14 days prior to the first dose of study drugs
6. Anticoagulant or thrombolytic agent within 10 days prior to the first dose of study drugs.
7. Evidence and history of severe bleeding tendency or coagulation dysfunction.
8. The toxicity of previous anti-tumor therapy has not been alleviated.
9. Symptomatic central nervous system metastases (CNS) metastasis and/or cancerous meningitis.
10. Have suffered from the second primary active malignant tumor in the past 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 2 years
  Objective response rate is the proportion of subjects with complete response (CR) or partial response (PR), based on RECIST v1.1.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to approximately 2 years
  Progression free survival is defined as the time from the start of treatment until the first documentation of disease progression or death due to any cause, whichever occurs first (based on RECIST v1.1).
Overall survival (OS) | Up to approximately 2 years
  OS is the time from the date of randomization or first dosing date to death due to any cause.
Disease control rate (DCR) | Up to approximately 2 years
  DCR is defined as the proportion of subjects with CR, PR, or stable disease(SD) based on RECIST v1.1.
Duration of response (DoR) | Up to approximately 2 years
  DoR is defined as the duration from the first documentation of objective response to the first documented disease progression (based on RECIST v1.1) or death due to any cause, whichever occurs first.
Time to response (TTR) | Up to approximately 2 years
  TTR is defined as the time from the start of the treatment to the first objective tumor response observed for patients who achieve CR or PR (based on RECIST v1.1).
Pharmacokinetic (PK) parameters | Up to 30 days after last treatment
  The PK parameters include serum concentrations of PM8002 at different timepoints after study drug administration.
Anti-drug antibody(ADA) | Up to 30 days after last treatment
  To evaluate the incidence of ADA to PM8002
Treatment related adverse events (TRAEs) | Up to 30 days after last treatment
  The incidence and severity of TRAEs graded according to NCI-CTCAE v5.0
Correlation between PD-L1 expression and antitumor effect | Up to approximately 2 years
  To evaluate correlation between PD-L1 expression and antitumor effect

OTHER OUTCOMES:
Population PK analysis | Up to 30 days after last treatment
  To assess the Exposure-Response of PM8002 by means of population PK (popPK) analysis
Correlation between PM8002 exposure, immunogenicity and efficacy | Up to approximately 2 years
  To evaluate correlation between PM8002 exposure, immunogenicity and efficacy
Correlation between PM8002 exposure, immunogenicity and safety | Up to 30 days after last treatment
  To evaluate correlation between PM8002 exposure, immunogenicity and safety

CONTACTS AND LOCATIONS:
Overall Officials: Wu Yilong, PhD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Medical Ethics Committee of Guangdong Provincial People's Hospital, Guangzhou, Guangdonng, China

IPD SHARING:
Plan to Share IPD: Yes
The data will be published or presented for publications (poster, abstract, articles or papers) or any presentations.
Time Frame: After the trial completed
Access Criteria: NCI is committed to sharing data in accordance with NIH policy.